CLINICAL TRIAL: NCT00256555
Title: GROWTH HORMONE USE IN CYSTIC FIBROSIS - A MULTICENTER STUDY
Brief Title: Growth Hormone Treatment Study in Children With Cystic Fibrosis
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 999-M02
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Growth Hormone

STUDY DESIGN:
Intervention Model Description: 00

INTERVENTIONS:
Drug: Nutropin AQ

SUMMARY:
Cystic fibrosis (CF) is a catabolic condition, and children affected with this disease frequently have problems with growth, despite adequate nutrition. We hypothesize that the anabolic effects of growth hormone (GH) will improve the height and weight of CF patients and thereby improve their clinical status and their quality of life. We further hypothesize that these effects will be sustained for at least one year after GH treatment is complete.

DETAILED DESCRIPTION:
We will test our hypotheses by recruiting 40 CF children from five CF centers (8 per center) across the country. Patients will be randomly assigned to receive treatment with GH (0.3 mg/kg/wk) during the first 12 months, or during the second 12 months. All subjects will be followed every three months for the entire 24 months. Growth data and PFT data from the year prior to study will be obtained from the medical record for each subject. Our specific aims include:

1. To determine the effect of GH on height, height velocity, body weight and lean body mass. We will measure height and weight using a standardized stadiometer and scale, respectively, every three months during the study. From these measurements we will calculate height and weight velocity and height and weight Z score. Lean body mass (LBM) will be measured by DEXA every six months. Baseline height and weight will be analyzed as covariates to determine whether children whose height and/or weight are at the lowest percentiles achieve greater improvement in height and weight velocity and lean body mass. This specific aim tests the hypothesis that GH significantly improves height, height velocity, weight, weight velocity and lean body mass in CF children irrespective of growth prior to starting the drug.
2. To determine the effect of GH on pulmonary function. Pulmonary function tests, including FEV1, FVC and PImax and PEmax (for estimation of respiratory muscle strength), will be measured at baseline and every 6 months in all subjects. We will document inpatient admissions and outpatient antibiotic therapy during the study. Baseline pulmonary function will be analyzed as a covariate to determine whether children with good pulmonary function achieve greater benefit than children with poor pulmonary function. This specific aim tests the hypothesis that GH use improves pulmonary function in CF children regardless of level of pulmonary functions prior to using the drug.
3. To determine if GH use in CF patients positively impacts quality of life. At baseline and every six months, we will administer a 15 minute questionnaire to both the parent and patient to assess quality of life. These questionnaires entitled "The Cystic Fibrosis Questionnaire" have been recently developed and tested for quality. They are specific for CF patients and have been approved by the National CF Foundation. This specific aim will test the hypothesis that GH use improves quality of life in CF patients.
4. To determine if the clinical improvement obtained from GH use is sustained. Those patients treated with GH during the first 12 months will be followed for 12 months after treatment to determine if the outcome variables remain better than baseline after growth hormone therapy is discontinued. This specific aim tests the hypothesis that GH use results in sustained improvement in height velocity, weight velocity, lean body mass, pulmonary function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* prepubertal CF patients (ages 5-12)
* capable of performing pulmonary function tests
* less than the 25th percentile for age and sex normal values for height and/or weight.

Exclusion Criteria:

* previous diagnosis with diabetes
* previous insulin requirement
* inability to perform pulmonary function testing
* colonization with burkholderia cepacia

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2000-02 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana S. Hardin, M.D., Principal Investigator — University of Texas Southwestern Medical Center

REFERENCES:
- [Background] Hardin DS. GH improves growth and clinical status in children with cystic fibrosis -- a review of published studies. Eur J Endocrinol. 2004 Aug;151 Suppl 1:S81-5. doi: 10.1530/eje.0.151s081. PMID 15339250
- [Background] Hardin DS. Growth hormone treatment in children with cystic fibrosis. Minerva Pediatr. 2002 Oct;54(5):365-71. PMID 12244275
- [Background] Hardin DS. Growth problems and growth hormone treatment in children with cystic fibrosis. J Pediatr Endocrinol Metab. 2002 May;15 Suppl 2:731-5. PMID 12092687
- [Background] Hardin DS, Ellis KJ, Dyson M, Rice J, McConnell R, Seilheimer DK. Growth hormone improves clinical status in prepubertal children with cystic fibrosis: results of a randomized controlled trial. J Pediatr. 2001 Nov;139(5):636-42. doi: 10.1067/mpd.2001.117578. PMID 11713439
- [Background] Hardin DS, Ellis KJ, Dyson M, Rice J, McConnell R, Seilheimer DK. Growth hormone decreases protein catabolism in children with cystic fibrosis. J Clin Endocrinol Metab. 2001 Sep;86(9):4424-8. doi: 10.1210/jcem.86.9.7822. PMID 11549686
- [Result] Hardin DS, Rice J, Ahn C, Ferkol T, Howenstine M, Spears S, Prestidge C, Seilheimer DK, Shepherd R. Growth hormone treatment enhances nutrition and growth in children with cystic fibrosis receiving enteral nutrition. J Pediatr. 2005 Mar;146(3):324-8. doi: 10.1016/j.jpeds.2004.10.037. PMID 15756212